CLINICAL TRIAL: NCT02440607
Title: The Effect of an Electronic Dynamic Cognitive Aid Versus a Static Cognitive Aid on the Management of a Simulated Crisis
Brief Title: Effect of an Electronic Cognitive Aid Versus Static Cognitive Aid on the Management of a Simulated Crisis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EH15-111
Record Dates: First submitted 2015-04-22; First posted 2015-05-12 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Cognitive Aids
Keywords: Randomization; cognitive aids types; aids
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic aid (Experimental): The dynamic aid will consist of a centralized electronic aid embedded within a simulated EMR.
  Interventions: Other: Electronic Cognitive Aid
- Static Cognitive aid (Active Comparator): The static aid represents the standard algorithm put forth by a leading clinical care organization.
  Interventions: Other: Static Cognitive Aid

INTERVENTIONS:
Other: Electronic Cognitive Aid
  Arms: Electronic aid
Other: Static Cognitive Aid
  Arms: Static Cognitive aid

SUMMARY:
Clinical decision support tools with in the electronic medical record can improve clinical care processes. To date, there is little evidence evaluating crisis management with such decision support tools. The investigators aim to create an electronic cognitive aid with embedded decision support to aid clinicians during the management of a crisis. In order to test the effectiveness of this tool, investigators seek to compare the simulated medical management of a crisis (malignant hyperthermia) using a traditional cognitive aid (laminated card) versus a dynamic electronic visual aid with decision support.

ELIGIBILITY:
Inclusion Criteria:

* resident physicians training in Anesthesia

Exclusion Criteria:

* Non resident anesthesia providers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Performance on Task Checklist | Time 0-30min
  Number of tasks successfully performed as rated on video review
Anesthesia Nontechnical skills score | Time0-30min
  Overall performance score; Video of management of crisis will be reviewed after completion of the scenario.

CONTACTS AND LOCATIONS:
Locations (1):
- Grainger Center for Simulation, Evanston, Illinois, United States

REFERENCES:
- [Derived] Shear TD, Deshur M, Benson J, Houg S, Wang C, Katz J, Aitchison P, Ochoa P, Wang E, Szokol J. The Effect of an Electronic Dynamic Cognitive Aid Versus a Static Cognitive Aid on the Management of a Simulated Crisis: A Randomized Controlled Trial. J Med Syst. 2018 Nov 22;43(1):6. doi: 10.1007/s10916-018-1118-z. PMID 30467609